CLINICAL TRIAL: NCT03173053
Title: Long-term StaphyloCoccus Aureus decolonizAtion in Patients on Home parenteRal nutRition: a randomIzed multicEnter tRial.
Brief Title: S. Aureus Decolonization in HPN Patients.
Acronym: CARRIER
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Results interim-analysis
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NL 61885.091.17
Record Dates: First submitted 2017-05-29; First posted 2017-06-01 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2020-10

CONDITIONS: Staphylococcus Aureus; Motility Disorder
Keywords: S. aureus; Home Parenteral Nutrition; Intestinal failure; Eradication; Decolonization
MeSH Terms: conditions — Staphylococcal Infections; Intestinal Failure | interventions — Doxycycline; Trimethoprim; Trimethoprim, Sulfamethoxazole Drug Combination; Clindamycin; Clarithromycin; Ciprofloxacin; Fusidic Acid; Rifampin; Chlorhexidine; Mupirocin; Povidone-Iodine

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized controlled, open label superiority trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Search and destroy (SD) strategy (Active Comparator): A quick and, short topical decolonization treatment combined with systemic antibiotics for S. aureus.
  Drug: Doxycycline 200mg once daily during one week Drug: Trimethoprim 200mg twice daily during one week Drug: Co-trimoxazol (Sulfamethoxazole/trimethoprim) 960mg twice daily during one week Drug: Clindamycin 600mg thrice daily during one week Drug: Clarithromycin 500mg twice daily during one week Drug: Ciprofloxacin 750mg twice daily during one week Drug: Fusidic acid (tablet) 500mg thrice daily during one week Drug: Rifampin 600mg twice daily during one week Drug: Mupirocin nasal ointment 20mg/g thrice daily during one week Drug: Fusidic acid ointment 20mg/g thrice daily during during five days Drug: Chlorhexidine body wash 40 mg/ml once daily during five days Drug: Betadine shampoo 75 mg/ml once daily during five days Drug: Chlorhexidine oropharyngeal rinse 2mg/ml thrice daily during five days
  Interventions: Drug: Doxycycline; Drug: Trimethoprim; Drug: Sulfamethoxazole/trimethoprim; Drug: Clindamycin; Drug: Clarithromycin; Drug: Ciprofloxacin; Drug: Fusidic Acid; Drug: Rifampin; Drug: Chlorhexidine; Drug: Mupirocin; Drug: Betadine
- Continuous suppression (CS) strategy (Active Comparator): A repeated, continuous, topical decolonization treatment of S. aureus
  Drug: Mupirocin nasal ointment 20mg/g thrice daily during one week Drug: Fusidic acid ointment 20mg/g thrice daily during during five days Drug: Chlorhexidine body wash 40 mg/ml once daily during five days Drug: Betadine shampoo 75 mg/ml once daily during five days Drug: Chlorhexidine oropharyngeal rinse 2mg/ml thrice daily during five days
  Interventions: Drug: Chlorhexidine; Drug: Mupirocin; Drug: Betadine

INTERVENTIONS:
Drug: Doxycycline — tablet
  Arms: Search and destroy (SD) strategy
Drug: Trimethoprim — tablet
  Arms: Search and destroy (SD) strategy
Drug: Sulfamethoxazole/trimethoprim — tablet
  Other Names: Bactrimel
  Arms: Search and destroy (SD) strategy
Drug: Clindamycin — tablet
  Arms: Search and destroy (SD) strategy
Drug: Clarithromycin — tablet
  Arms: Search and destroy (SD) strategy
Drug: Ciprofloxacin — tablet
  Arms: Search and destroy (SD) strategy
Drug: Fusidic Acid — tablet or ointment
  Arms: Search and destroy (SD) strategy
Drug: Rifampin — tablet
  Arms: Search and destroy (SD) strategy
Drug: Chlorhexidine — Mouthwash or bodywash
Drug: Mupirocin — Nasal ointment
Drug: Betadine — Shampoo

SUMMARY:
This trial focusses on identifying the most effective and safe long-term S. aureus carriage decolonization strategy in home parenteral nutrition patients. Half of the participants will receive a quick and short systemic antibiotic treatment combined with topical treatment, while the other half will receive only topical treatment on a periodic basis.

DETAILED DESCRIPTION:
Patients on home parenteral nutrition (HPN) are exposed to a lifelong risk of developing S. aureus bacteremia (SAB). SAB pose a threat to both catheter and patient survival and may lead to a permanent loss of vascular access. S. aureus carriage eradication has proven successful in prevention of S. aureus infections. S. aureus decolonization is a key strategy to maintain venous access and avoid hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Patient is fully able to understand the nature of the proposed intervention.
* Written informed consent by the patient before entering the trial.
* Age ≥ 18 years.
* Estimated life expectancy ≥ 1 year.
* Patient colonized with S. aureus.

Exclusion Criteria:

* Cannot be expected to comply with the trial plan (substance abuse, mental condition).
* Pregnant or breastfeeding women.
* Continuous exposure to Methicillin-resistant S. aureus (MRSA; e.g. pig farmer).
* Allergy for chlorhexidine and betadine.
* No options for oral and/or topical antibiotics due to allergies.
* Active S. aureus infection.
* Currently on treatment with antibiotics active against S. aureus.
* Decolonization (including mupirocin) treatment in the previous two months.
* The presence of a nasal foreign body.
* Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) levels more than five times the upper limit of normal or liver failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2021-10-14 (Actual); Study Completion 2021-10-14 (Actual)

PRIMARY OUTCOMES:
Proportion of patients totally eradicated for S. aureus during one year | One year
  Totally eradicated is defined as 100% of all culture swabs (nose, throat, rectum), exit-site catheter and body regions on indication) being negative for S. aureus.

SECONDARY OUTCOMES:
Proportion of patients totally eradicated after one year | One year
  Proportion of patients totally eradicated for S. aureus based on negative cultures performed after one year
Developing long-term antimicrobial resistance | 6 and 12 months
  Long-term antimicrobial resistance at 6 and 12 months (measured with standard cultures and NGS)
Incidence of S. aureus infections | Every 3 months during one year
  Incidence of S. aureus infections measured with (serious) adverse events forms every 3 months
Overall incidence of infections | Every three months during one year
  Overall incidence and time to onset of infections measured with (serious) adverse events forms every 3 months
Number of catheter removals | One year
  Number of catheter removals based on data from electronic patient dossier
Mortality | One year
  Mortality based on data from electronic patient dossier
S. aureus transmission | One year
  S. aureus transmission routes from caregiver to patient (measured with NGS).
Patient compliance | Every three months during one year
  Patient compliance (measured with medication files, counting pills, trial-specific medication diary).
Adverse events | Every three months during one year
  Adverse events (measured with (serious) adverse event forms every 3 months).
Predictors for infections and treatment outcome | One year
  Predictors for infections and treatment failure/success (binominal regression analysis).
Health related quality of life | 0, 6 and 12 months
  Generic health related quality of life (measured with a validated questionnaire (EQ5D-5L)).
Healthcare related costs. | One year
  Cost-effectiveness analysis

CONTACTS AND LOCATIONS:
Overall Officials: Joost PH Drenth, MD, PhD, Study Director — Sponsor GmbH
Locations (4):
- Denmark (2):
  - Aalborg Universitetshospital, Aalborg
  - Rigshospitalet, Copenhagen
- Netherlands (2):
  - Radboud UMC, Nijmegen, Gelderland
  - AMC, Amsterdam, North Holland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gompelman M, Wezendonk GTJ, Wouters Y, Beurskens-Meijerink J, Fragkos KC, Rahman FZ, Coolen JPM, van Weerdenburg IJM, Wertheim HFL, Kievit W, Akkermans RP, Serlie MJ, Bleeker-Rovers CP, Wanten GJA. Randomized clinical trial: Long-term Staphylococcus aureus decolonization in patients on home parenteral nutrition. Clin Nutr. 2023 May;42(5):706-716. doi: 10.1016/j.clnu.2023.03.010. Epub 2023 Mar 17. PMID 36965196
- [Derived] Gompelman M, Wouters Y, Kievit W, Hopman J, Wertheim HF, Bleeker-Rovers CP, Wanten GJA. Long-term Staphylococcus aureus decolonization in patients on home parenteral nutrition: study protocol for a randomized multicenter trial. Trials. 2018 Jun 28;19(1):346. doi: 10.1186/s13063-018-2732-2. PMID 29954418